<u>Official Title</u>: A Prospective, Multicentre, Open Clinical Investigation Evaluating Clinical Performance, Safety and Patient Reported Outcomes With an Active Osseointegrated Steady-State Implant System (OSI) in Adult Subjects With Conductive Hearing Loss, Mixed Hearing Loss or Single-sided Sensorineural Deafness

NCT Number: NCT04041700

**Document Date**: 26 March 2020



# Statistical Analysis Plan

Clinical Investigation Title:

A prospective, multicentre, open clinical investigation evaluating clinical performance, safety and patient reported outcomes with an Active Osseointegrated

Stoody State Implent System (OSI) in adult subjects with

Steady-State Implant System (OSI) in adult subjects with conductive hearing loss, mixed hearing loss or single-

sided sensorineural deafness.

Clinical Investigation Short Title: Clinical performance, safety and PROs of an Active

Osseointegrated Steady-State Implant System (OSI)

Clinical Investigation Number: CBAS5751

**Related CIP:** D1622635, 2.0

Clinical Project Manager (CPM):

Cochlear Bone Anchored Solutions AB

Konstruktionsvägen 14

PO Box 82

Mölnlycke, Sweden, SE-435 22

Statistical Analysis Plan author/s:

Statistiska konsultgruppen

SAP Version: 1.0

Date: 26-MAR-2020

# Contents

| 1 | Introd | uction | | 3 |
|---|---|---|---|---|
| | 1.1 | Schedu | le of events | 3 |
| 2 | Study | populati | on | 5 |
| 3 | Statis | tics | | 5 |
| | 3.1 | Sample | Size | 5 |
| | 3.2 | Analyse | s | 6 |
| | | 3.2.1 | Pass/Fail Criteria | 6 |
| | | 3.2.2 | Hypotheses | 6 |
| | | 3.2.3 | Primary Hypotheses | 6 |
| | | 3.2.4 | Secondary Hypotheses | 7 |
| | | 3.2.5 | Additional statistical issues | 8 |
| | 3.3 | Analysis | s Datasets | 9 |
| | | 3.3.1 | Safety | 9 |
| | | 3.3.2 | Intent-to-Treat | 9 |
| | | 3.3.3 | Per Protocol dataset | 9 |
| | 3.4 | Addition | al Statistical Considerations | 9 |
| | | 3.4.1 | Missing, Unused or Spurious Data | 9 |
| | | 3.4.2 | Planned Interim Analysis | 10 |
| | | 3.4.3 | Criteria for Termination of the Clinical Investigation | 10 |
| | | 3.4.4 | Additional Statistical Analyses | 10 |
| | 3.5 | Conduc | t of Statistical Analysis | 13 |
| | | 3.5.1 | Timing of analyses | 13 |
| | 3.6 | Quality | control on statistical analysis | 14 |
| | 3.7 | Present | ation of data | 14 |
| | | 3.7.1 | General | 14 |
| | | 3.7.2 | List of tables | 14 |
| | | 3.7.3 | List of figures | 16 |
| 4 | Refer | ences | | 17 |
| | 4.1 | Internal | References | 17 |
| | 4.2 | Externa | l References | 17 |
| 5 | Chan | ge Histor | у | 17 |
| 6 | Defini | tions | | 17 |



#### 1 INTRODUCTION

This document is a companion document to the Clinical Investigation Plan (CBAS5751). It includes a comprehensive description of the sample size estimation, the intended statistical analyses with reference to the primary and secondary hypotheses, and additional statistical considerations such as the intended treatment of missing data.

Any deviation from the Statistical Analysis Plan will be reported in the Clinical Investigation Report.

#### 1.1 Schedule of events

| | Screening<br>And<br>Baseline | Surgery | Suture<br>removal | Fitting | Follow up<br>6W | Follow up<br>3M | Follow up<br>6M |
|---|---|---|---|---|---|---|---|
| Timing of visit | | 0 | 2W | 4W | 6W | 3M | 6M |
| Visit window (±) | | | ±5D | ±1W | ± 1W | ± 2W | ± 3W |
| Procedures | | | | | | | |
| Written informed consent | х | | | | | | |
| Demographics | Х | | | | | | |
| Eligibility | Х | | | | | | |
| Medical history | Х | | | | | | |
| Hearing history | X | | | | | | |
| Device history | Х | | | | | | |
| Audiogram | Xa | | | | | | |
| Soft tissue thickness | x | 3 | | | | | |
| Surgery | | Xp | | | | | |
| Suture removal | | | X | | | | |
| Sound processor fitting | Xc | | | х | Xq | Xq | Xq |
| Microphone placement | | | | X | | | |
| Fine tuning | | | | Х | Xq | Xq | Xq |
| Feedback<br>measurements | | | | Х | Xe | Xe | Xe |
| Coil-to-coil measurements | | | | х | Xe | Xe | Xe |
| BC Direct | Xf | | | Х | Xe | Xe | Xe |
| Free field<br>thresholds | X <sup>f, g</sup> | | | Х | | х | х |
| Speech recognition in quiet | X <sup>f, g</sup> | | | Х | | х | Х |
| Speech recognition in noise | X <sup>f, g, h</sup> | | | Х | | Х | х |
| APHAB | Χg | | | | | X | X |

| | Screening<br>And<br>Baseline | Surgery | Suture<br>removal | Fitting | Follow up<br>6W | Follow up<br>3M | Follow up<br>6M |
|---|---|---|---|---|---|---|---|
| Timing of visit | | 0 | 2W | 4W | 6W | 3M | 6M |
| Visit window (±) | | | ±5D | ±1W | ± 1W | ± 2W | ± 3W |
| SSQ | Xg | | | | | Х | X |
| HUI | Xh | | | | | Х | Х |
| Usability | | | | Xi | Xi | Xi | Xi |
| Numbness | | | X | X | X | Х | X |
| Device exposure j | | Х | X | Х | X | X | Х |
| Adverse Events | X | X | X | X | X | Х | X |
| Device Deficiencies | | X | | X | X | Х | Х |
| Concomitant therapies | х | Х | х | х | Х | X | х |
| Extra visits as needed | | | | | | | |

Abbreviations: BC, Bone Conduction; APHAB, Abbreviated Profile of Hearing Aid Benefit; SSQ, Speech, Spatial and Qualities of Hearing Scale; HUI, Health Utilities Index

<sup>i</sup>Usability: Magnet choice, Sound Processor retention, Sound Processor wearing comfort at first fitting and all follow up visits, Daily use, Daily streaming, Battery life time, Use of SoftWear pad at all follow up visits.

<sup>j</sup> "Device exposure" is to collect information about for how long the subject is exposed to the Osia 2 Sound Processor and Osia 2 Implant. Data is summarized from other case report form pages.

<sup>&</sup>lt;sup>a</sup> An audiogram not older than 6 months can be used if it contains all the required frequencies (250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000Hz).

<sup>&</sup>lt;sup>b</sup>Surgical variables: Surgery time, Bone polishing/removal at the actuator site, Bl300 Implant length, Location of Bl300 Implant, Type of anesthesia, Soft tissue reduction, Surgical incision type, Length of the surgical incision, Placement of the coil, Soft tissue thickenss, Location of surgical incision

<sup>&</sup>lt;sup>c</sup>Should be performed with Baha 5 Power at Screening and Baseline

dShould be done if needed.

<sup>&</sup>lt;sup>e</sup> Should be performed at each occasion the software is being used to fit or fine tune the device <sup>f</sup>Baha 5 Power Sound Processor on Baha Softband.

<sup>&</sup>lt;sup>g</sup> Unaided.

hIn a preoperative hearing situation



#### 2 STUDY POPULATION

The rationale for conducting this clinical investigation is to gather clinical data on patients implanted with the OSI200 Implant. While the non-clinical and clinical data all indicate that the Osia 2 System will perform as intended and provide a bone conduction hearing implant (BCHI) system with a similar, or improved, safety profile as its CE-marked predecessor device, which is currently being used by more than one hundred recipients world-wide, it is of utmost interest to assess the performance and safety of the Osia 2 System when used as intended.

The following sites will be participating in the study.

| Site | Planned number of patients |
|---|---|
| The Royal Victorian Eye and Ear Hospital | 10-15 |
| Sydney Cochlear Implant Centre | 10-15 |
| Department of Otorhinolaryngology, Head and Neck Surgery, Faculty of Medicine, The Chinese University of Hong Kong | 10-15 |

Subgroup analyses will also be performed on one group consisting of Mixed/conductive subjects and one consisting of SSD subjects.

#### 3 STATISTICS

### 3.1 Sample Size

Based on 6 months safety data from 51 subjects implanted with the predecessor Osia System at 5 clinics in the multicentre clinical investigation described in section 4.2.2.1 it is judged that approximately 10 subjects per clinic and 3 clinics is reasonable for detecting any safety issues with the Investigational device in this study. The primary safety evaluation will be performed 3 months post-surgery, which with an estimation of 30 subjects will equate 7.5 patient years. This is considered to be enough safety data for the primary safety analysis.

With a total of 30 subjects, there will be a very high power to detect significant changes in the primary performance evaluations audiometric thresholds (PTA4) and adaptive speech in noise (speech to noise ratio, SNR) at 3 months.

PTA4: Assuming the same mean reduction in PTA4 as in the multicentre clinical investigation of the predecessor Osia System (Mean change -25 dB, SD 9.5 dB), the resulting power with 30 subjects is 0.99.

SNR: In the multicentre clinical investigation of the predecessor Osia System a change in SNR from 4.98 dB (SD 7.76 dB) unaided to -8.19 dB (SD 6.58 dB) aided resulted in a mean improvement in SNR of -13.3 dB (SD 8.1 dB). In that investigation, speech was presented from the front and noise from the rear speaker. In the present investigation, however, both speech and noise will be presented from the front speaker, which is known to result in higher SNR values in the aided situation (the SNR in the unaided situation is not expected to change significantly). In a pilot clinical investigation conducted at Cochlear's own research facility (CBAS5271, Sub study 118), a mean SNR value of -2.5 dB was recorded

with the Investigational device (Osia 2 System). Assuming that in the present investigation the unaided mean SNR is similar to the unaided scores in the multicenter investigation and that the aided mean SNR is similar to the pilot investigation, a mean improvement in SNR of approximately -7.6 dB (SD 8.1 dB) is expected. With 30 subjects, the resulting power is 0.99.

## 3.2 Analyses

#### 3.2.1 Pass/Fail Criteria

Not Applicable.

#### 3.2.2 Hypotheses

The hierarchical testing procedure below is introduced to guarantee that the probability of Type I error is < 5% for all confirmative statements. The order of the hierarchical testing procedure will be:

- 1. PTA 4 pre-operative unaided vs. 3 months post-surgery (Primary efficacy analysis)
- 2. Adaptive speech recognition in noise (50% performance), signal to noise ratio (SNR) pre-operative unaided vs. 3 months post-surgery
- 3. Speech in quiet at 65dB SPL pre-operative unaided vs. 3 months post-surgery
- 4. APHAB Global pre-operative unaided vs. 3 months post-surgery
- 5. Hearing attribute (HUI) pre-operative situation vs. 3 months post-surgery
- Mean of the 12 items (Total score) in the SSQ pre-op unaided vs. 3 months postsurgery

If the first analysis is significant the probability mass 0.05 will go to the second analysis. If the second analysis is also significant the probability mass 0.05 will go to the third analysis and so on. When the first non-significant analysis is reached this and all analyses thereafter will be non-confirmative while the previous analyses will be confirmative. If the first analysis is non-significant no analysis will be confirmative. All testing will be Alpha level of 0.05 and two-sided test will be used and the analysis will be performed on the ITT.

#### 3.2.3 Primary Hypotheses

Group mean free-field PTA4 (average of 500, 1000, 2000, and 4000 Hz) with the Investigational device at the 3-month postoperative interval will be improved over that measured preoperatively in the unaided condition (baseline).

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 = 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 \neq 0$ .

where:

 $\alpha_0$  = baseline preoperative PTA4;

 $\mu_F$  = mean follow-up PTA4 3 months postoperative.

# Cooklean

# **CBAS Master template (Word)**

Change in free-field threshold audiometry: PTA4 (mean of 500, 1000, 2000 and 4000Hz), from unaided versus Investigational device at 3 months post-surgery visit for the ITT population, using Fisher's two-sided non-parametric permutation test for paired observations to demonstrate an improvement in PTA4.

Alpha level of 0.05 and two sided test will be used and the analysis will be performed on the ITT population.

Group mean Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR) with the Investigational device at the 3-month postoperative interval will be improved over that measured preoperatively in the unaided condition.

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 = 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 \neq 0$ ,

where:

 $\alpha_0$  = baseline preoperative Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR);

 $\mu_F$  = mean follow-up Adaptive speech recognition in noise (50% performance), speech to noise ratio (SNR) 3 months postoperative.

Change in Adaptive speech recognition in noise (50% performance), from unaided versus Investigational device at 3 months post-surgery visit for the ITT population, using Fisher's two-sided non-parametric permutation test for paired observations to demonstrate an improvement in PTA4.

Alpha level of 0.05 and two sided test will be used and the analysis will be performed on the ITT population.

Both PTA4 and SNR must be significant at alpha 0.05 for the primary analysis to be considered as confirmative.

Missing data will be handled according to 3.4.1.

#### 3.2.4 Secondary Hypotheses

Group mean **Speech in quiet at 65dB** when using the Investigational device at 3 months postoperative compared to the unaided hearing using Fisher's two-sided non-parametric permutation test for paired observations.

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 = 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 \neq 0$ ,

where:

 $\alpha_0$  = baseline preoperative word recognition score;

 $\mu_F$  = mean follow-up word recognition score 3 months postoperative.

Group mean Global score using the Abbreviated Profile of Hearing Aid Benefit (APHAB) when using the Investigational device at 3 months post surgery compared to

unaided hearing, using Fisher's two-sided non-parametric permutation test for paired observations.

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 = 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 \neq 0$ ,

where:

 $\alpha_0$  = baseline APHAB Global score;

 $\mu_F$  = mean follow-up APHAB Global score 3 months postoperative.

Group mean **Hearing attribute (HUI)** when using the Investigational device at 3 months post surgery compared to the preoperative hearing situation, using Fisher's two-sided non-parametric permutation test for paired observations.

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 = 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 \neq 0$ ,

where:

 $\alpha_0$  = baseline Hearing attribute (HUI);

 $\mu_F$  = mean follow-up Hearing attribute (HUI) 3 months post-fitting.

Group mean Total score using the Speech, Spatial and Qualities of Hearing Scale (SSQ) when using the Investigational device at 3 months post surgery compared to the unaided hearing, using Fisher's two-sided non-parametric permutation test for paired observations.

This endpoint is represented by the following hypotheses:

$$H_0$$
:  $\mu_F - \alpha_0 = 0$ ,

$$H_a$$
:  $\mu_F - \alpha_0 \neq 0$ ,

where:

 $\alpha_0$  = baseline SSQ Total score;

 $\mu_F$  = mean follow-up SSQ Total score 2 months post-fitting.

Missing data will be handled according to 3.4.1.

All other secondary outcomes will not be formally hypothesis tested but summarized and p-values will be calculated.

In addition to comparing follow up data with unaided analyses will also be made with Baha Power sound processor on a Baha Softband (screening).

#### 3.2.5 Additional statistical issues

If any paired analysis of dichotomous and ordered categorical variables (i.e. if any continuous variables will be categorized) will be made the Sign test will be used.



The main efficacy analyses will be performed at 3 months after surgery on the ITT population and complementary efficacy analyses will be performed 6 months after surgery on the ITT population. In addition, all analyses will be made on the PP population. Sub analyses will also be performed on one group consisting of Mixed/conductive subjects and one consisting of SSD subjects.

Primary safety analysis will be performed at 3 months post-surgery.

### 3.3 Analysis Datasets

The final definition of the analysis sets (ITT, PP and Safety) will be taken at the clean file meeting before database lock.

All efficacy analyses will be performed on both ITT and PP populations.

#### 3.3.1 **Safety**

The Safety population/dataset consists of all surgically treated subjects.

#### 3.3.2 Intent-to-Treat

The Intention-to-Treat population/dataset (ITT) will include all subjects who have undergone surgical intervention.

Missing data will be handled according to 3.4.1.

#### 3.3.3 Per Protocol dataset

The Per Protocol population/dataset (PP) will include subjects that have completed the study according to the protocol. Subjects that were incorrectly included or were considered major protocol violators that affect the primary analysis should be removed from the PP population/dataset.

Missing data will be handled according to 3.4.1.

#### 3.4 Additional Statistical Considerations

#### 3.4.1 Missing, Unused or Spurious Data

All ITT analyses will be performed/presented both for the imputed (main analyses) and for the non-imputed data (sensitivity analyses).

Imputation of missing values will be performed for all efficacy variables. No imputation of baseline values or baseline carry forward will be made. Imputations will be made according to the following rules:

- If a value is missing at the end of a time period for a patient, last observation will be carried forward.
- If a missing value is occurring between two time points with values, an interpolation will be made for continuous variables and for categorical variables the value from the previous visit will be carried forward.
- 3. As a sensitivity analysis imputation of missing values will be performed for all efficacy variables using stochastic regression imputations.

Spurious data will be cleaned prior to clean file meeting. If spurious data are detected after clean file is declared actions to consider will be;

- 1. unlock, correction of the spurious data and a new re-lock will be made alternatively,
- 2. a sensitivity analysis will be performed that accounts for the spurious data in a proper statistical fashion (e.g. non parametric methods).

### 3.4.2 Planned Interim Analysis

No interim analyses are planned to be performed.

#### 3.4.3 Criteria for Termination of the Clinical Investigation

Not applicable.

#### 3.4.4 Additional Statistical Analyses

#### 3.4.4.1 Major protocol deviations

Major protocol deviations are those that are considered to have an effect on the analysis. The number of patients with major protocol deviations will be summarised per treatment group. A list of protocol deviations will be produced.

#### 3.4.4.2 Demographics

A descriptive presentation of demographic data will be presented as described in paragraph 3.7:

- Age collected as date of birth (month and year)
- Gender
- Race
- Tobacco use
  - Never /Current/Former
  - Primary method (Cigarettes/Cigars/Pipe/eCigarettes/Chewing/Other)
  - Cigarettes/day

#### 3.4.4.3 Medical history

A descriptive presentation of medical history will be presented as described in paragraph 3.7:

- Relevant medical and surgical treatment during the past three years as judged by the investigator
- · Current concomitant medication and treatments

#### 3.4.4.4 Hearing history

Test ear (right/left)

A descriptive presentation of hearing history will be presented as described in paragraph 3.7:

- Type of hearing loss:
  - Conductive,
  - Mixed,
  - o SSD
- Aetiology of hearing loss:

# 00

# **CBAS Master template (Word)**

- o (chronic) infection,
- o tumour,
- o trauma.
- malformation,
- o otosclerosis,
- genetic
- unknown
- o other
- · History of hearing loss
  - o progressive
  - o progressive with sudden
  - sudden
  - congenital with progression (if age at onset was 0 month)
  - congenital without progression (if age at onset was 0 month)

#### 3.4.4.5 Device history

#### **Hearing aid**

- Has the subject used hearing aid (never/current/former)
- Has the subject used hearing aid (never/current/former) on test side
- Has the subject used hearing aid (never/current/former) on non-test side
   Has the subject used hearing aid (never/current/former) on both test side and non-test side

#### **Hearing Implant**

- Does the subject have and audiological implant (Never implanted/Implanted, still in use/Implanted, not in use/Explanted)
- Does the subject have and audiological implant (Never implanted/Implanted, still in use/Implanted, not in use/Explanted) on test side
- Does the subject have and audiological implant (Never implanted/Implanted, still in use/Implanted, not in use/Explanted) on non-test side
- Does the subject have and audiological implant (Never implanted/Implanted, still in use/Implanted, not in use/Explanted) on both test side and non-test side

All information collected in the eCRF regarding hearing aid and hearing implant will be listed.

#### 3.4.4.6 Audiogram

A descriptive presentation of audiograms at Screening will be presented (tabulated and graphically) as described in paragraph 3.7 by frequency (and Pure Tone Average (PTA4) for CHL and MHL (*mean of 500, 1000, 2000 and 4000Hz*) and for SSD (*mean of 500, 1000, 2000 and 3000Hz*)), test side, air/bone and masked/unmasked.

# 00

# **CBAS Master template (Word)**

#### 3.4.4.7 Soft tissue thickness

A descriptive presentation of Soft tissue thickness will be presented as described in paragraph 3.7.

#### 3.4.4.8 Surgery

A descriptive presentation of surgery data will be presented as described in paragraph 3.7:

- Treatment ear (indicate left or right or both. In case of both, indicate "test ear").
- Soft tissue thickness (mm)
- Type of anesthesia (general/local)
- Bone polishing/removal at the actuator site (yes/no)
- BI300 Implant length (3mm/4mm)
- Location of BI300 Implant (mm)
- Soft tissue reduction (yes/no)
- Surgical incision type (examples; C-shaped/S-shaped/straight)
- Location of the surgical incision in relation to the actuator (anterior/posterior)
- Estimated length of the surgical incision (mm)
- · Placement of the coil
  - o periosteal pocket (under periosteal)
  - o on top of periosteum
  - o on top of muscle
- Surgery time (time between first incision to last suture)

#### 3.4.4.9 Usability

A descriptive presentation of surgery data by visit will be presented as described in paragraph 3.7:

- Magnet choice
- Sound Processor retention
- Sound Processor wearing comfort
- Use of SoftWear pad
- Daily use
- Daily streaming
- Battery lifetime
  - Did the "low battery" signal occur (yes/no)

#### 3.4.4.10 BC Direct

A descriptive presentation of surgery data by visit will be presented as described in paragraph 3.7:

 BC Direct [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0 and 6.0 kHz] will be performed using a Baha Softband (preoperatively) at screening/baseline and using the Investigational device at fitting, 3- and 6-months post-surgery.

#### 3.4.4.11 Preoperative hearing aid

The difference in hearing performance at fitting- 3- and 6 months post-surgery when using the Investigational device compared to a preoperative hearing aid (if used by the patient) assessed as:

 The difference in Adaptive speech in noise [signal-to-noise ratio, 50% speech understanding].

#### 3.4.4.12 Coil-to-coil measurement

DLC measurements through-out the study will be presented.

#### 3.4.4.13 Implant site evaluation (numbness)

Implant site evaluation (numbness) will be summarised by frequency and percent of:

- No numbness,
- 2. Numbness over the implant Magnet Assembly area and
- Numbness over the implant Magnet Assembly area and 2 cm outside the implant Magnet Assembly area by visit.

#### 3.4.4.14 Adverse events

Separate tabulations of AEs, ADEs, SAEs, SADEs and AESIs will be produced. AEs, ADEs and AESIs will also be produced by severity (mild, moderate or severe) and relationship (related defined as Possibly, Probably and Definitely related). Number of events, number of subject and percent with events by System Organ Class (SOC, CTCAE) and CTCAE term will be presented.

#### 3.4.4.15 Device deficiency

DDs will be reported by visit as described in paragraph 3.7.

#### 3.4.4.16 Concomitant medication

Concomitant medications will be defined as start or end date from surgery to end of study and will be presented by listings.

### 3.5 Conduct of Statistical Analysis

The statistical analyses will be performed at Statistiska konsultgruppen by personnel employed at Statistiska konsultgruppen under supervision of the analyses will be performed by using SAS 9.4 (or later).

#### 3.5.1 Timing of analyses

The first reporting of analyses will be made when all patients have completed their 3 months visit of the data up to 3 months. This analysis is regarded as the primary analysis. At the end of the study, at 6 months, the second and final reporting of the study will be made including all data up to the 6 months visit including data prior to the 3 months visit (ie all data in the study).



# 3.6 Quality control on statistical analysis

Each programmer is responsible to continuously during working with data generation programs and statistical programs

#### 3.7 Presentation of data

#### 3.7.1 General

All data will be presented in summarized tables. The distribution of continuous variables as well as change in continuous variables will be given as n, mean, SD, SEM, Median, Min and Max and the distribution of dichotomous and categorical variables will be given as number and percentages. For continuous variables estimated mean and the 95% two-sided confidence interval (bootstrapped) for difference between groups will be presented. The hypotheses' p-values and the corresponding/accompanying estimated with a 95% Ci will be presented where applicable.

Selected variables will be presented in figures showing either box plots or mean (95% CI) over time on actual values and/or change. Audiogram data will be presented as traditional audiograms.

#### 3.7.2 List of tables

| Table | Title |
|---|---|
| Table 14.1.1 | Patient Disposition and Data Sets Analysed |
| | Protocol Deviations Leading to Exclusion from PP Population (ITT |
| Table 14.1.2 Population) | |
| Table 14.1.2.1 | Audiogram at screening - SSD patients (Safety Population) |
| Table 14.1.2.5 | Audiogram at screening - mixed/conductive patients (Safety Population) |
| Table 14.1.3.1 | Demographics and Baseline Characteristics (ITT Population) |
| Table 14.1.3.2 | Demographics and Baseline Characteristics (PP Population) |
| Table 14.1.4.1 | Device and hearing history (ITT Population) |
| Table 14.1.4.2 | Device and hearing history (PP Population) |
| Table 14.1.6 | Medical History (ITT Population) |
| Table 14.1.7 | Surgical History (ITT Population) |
| Table 14.1.8.1 | Prior Medications (ITT population) |
| Table 14.1.8.2 | Concomitant Medications (ITT population) |
| Table 14.1.9 Listing of Concomitant Treatments/Procedures (ITT population) | |
| Table 14.2.1.1 Threshold Audiometry - Free field Osia System vs Unaided (ITT Popula | |
| Table 14.2.1.2 Threshold Audiometry - Free field Osia System vs Unaided (PP Popula | |
| | Threshold Audiometry - Free field Osia System vs Unaided (landscape |
| Table 14.2.1.3 | layout) (All patients - ITT Population) |
| | Threshold Audiometry - Free field Osia System vs Unaided (landscape |
| Table 14.2.1.4 | layout) (Mixed/Conductive patients - ITT Population) |
| T 11 44045 | Threshold Audiometry - Free field Osia System vs Unaided (landscape |
| Table 14.2.1.5 | layout) (SSD patients - ITT Population) |
| T-LL- 44040 | Threshold Audiometry - Free field Osia System vs Unaided by Site (ITT |
| Table 14.2.1.6 Population) | |
| T-1-44047 | Threshold Audiometry - Free field (PTA-4) Osia System vs Unaided by Site |
| Table 14.2.1.7 | (ITT Population) |
| T-bl- 44004 | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.2.1 | Unaided (ITT Population) |



| 20 | · |
|---|---|
| Table 14.2.2.2 | Adaptive speech recognition in noise and Speech in quiet Osia System vs Unaided (PP Population) |
| 1 10 1000 0 10 1000 0 1 | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.2.3 | Unaided (landscape layout) (All patients - ITT Population) |
| Table 14.2.2.4 | Adaptive speech recognition in noise and Speech in quiet Osia System vs Unaided (landscape layout) (Mixed/Conductive patients - ITT Population) |
| 4 19 ANDERS NO MARKETON DE AMES | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.2.5 | Unaided (landscape layout) (SSD patients - ITT Population) |
| Table 14.2.2.6 | Adaptive speech recognition in noise and Speech in quiet Osia System vs Unaided by Site (ITT Population) |
| Table 14.2.2.7 | Listing of information regarding current hearing aid (ITT Population) |
| Table 14.2.3.1 | BC Direct (ITT Population) |
| Table 14.2.3.2 | BC Direct (PP Population) |
| Table 14.2.3.3 | BC Direct (landscape layout) (ITT Population) |
| Table 14.2.3.4 | BC Direct (landscape layout) (Mixed/Conductive patients - ITT Population) |
| Table 14.2.3.5 | BC Direct (landscape layout) (SSD patients - ITT Population) |
| Table 14.2.4.1 | HUI (ITT Population) |
| Table 14.2.4.2 | HUI (PP Population) |
| Table 14.2.4.3 | HUI (landscape layout) (ITT Population) |
| Table 14.2.4.4 | HUI (landscape layout) (HTT Population) HUI (landscape layout) (Mixed/Conductive patients - ITT Population) |
| 1(6) | |
| Table 14.2.4.5 | HUI (landscape layout) (SSD patients - ITT Population) |
| Table 14.2.5.1 | APHAB (ITT Population) |
| Table 14.2.5.2 | APHAB (PP Population) |
| Table 14.2.5.3 | APHAB (ITT Population) (landscape layout) (ITT Population) |
| Table 14.2.5.4 | APHAB (ITT Population) (landscape layout) (Mixed/Conductive patients - ITT Population) |
| Charles and the second of the | Expend (Contract and Annal Ann |
| Table 14.2.5.5 | APHAB (ITT Population) (landscape layout) (SSD patients - ITT Population) |
| Table 14.2.6.1 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (ITT Population) |
| Table 14.2.6.2 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (PP Population) The Speech, Spatial and Qualities of Hearing Scale (SSQ) (landscape layout) |
| Table 14.2.6.3 | (ITT Population) |
| Toble 14 0 C 4 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (landscape layout) |
| Table 14.2.6.4 | (Mixed/Conductive patients - ITT Population) |
| Table 14.2.6.5 | The Speech, Spatial and Qualities of Hearing Scale (SSQ) (landscape layout) (SSD patients - ITT Population) |
| Table 14.2.7.1 | Surgery (ITT population) |
| Table 14.2.7.2 | Surgery (PP population) |
| Table 14.2.8.1 | Usability (ITT population) |
| Table 14.2.8.2 | Usability (PP population) |
| Table 14.2.10.1 | Coil-to-coil measurement (ITT population) |
| Table 14.2.10.2 | Coil-to-coil measurement (PP population) |
| Table 14.2.10.1 | Threshold Audiometry - Free field Osia System vs Softband (ITT Population) |
| Table 14.2.10.2 | Threshold Audiometry - Free field Osia System vs Softband (PP Population) |
| | Threshold Audiometry - Free field Osia System vs Softband (landscape |
| Table 14.2.10.3 | layout) (All patients - ITT Population) |
| × | Threshold Audiometry - Free field Osia System vs Softband (landscape |
| Table 14.2.10.4 | |
| Table 14 0 40 5 | Threshold Audiometry - Free field Osia System vs Softband (landscape |
| Table 14.2.10.5 | layout) (SSD patients - ITT Population) |



| 20 | 78 |
|---|---|
| | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.11.1 | Softband (ITT Population) |
| | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.11.2 | Softband (PP Population) |
| | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.11.3 | Softband (landscape layout) (All patients - ITT Population) |
| | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.11.4 | Softband (landscape layout) (Mixed/Conductive patients - ITT Population) |
| | Adaptive speech recognition in noise and Speech in quiet Osia System vs |
| Table 14.2.11.5 | Softband (landscape layout) (SSD patients - ITT Population) |
| Table 14.3.1.1 | Summary of Adverse Events (Safety Population) |
| Table 14.3.1.2 | Adverse Events (AE), by CTCAE SOC and CTCAE Term (Safety Population) |
| | Adverse Device Events (ADE possibly, probably and definitely related), by |
| Table 14.3.1.3 | CTCAE SOC and CTCAE Term (Safety Population) |
| | Serious Adverse Events (SAE), by CTCAE SOC and CTCAE Term (Safety |
| Table 14.3.1.4 | Population) |
| | Adverse Events of Special Interest (AESI), by CTCAE SOC and CTCAE |
| Table 14.3.1.6 | Term (Safety Population) |
| Table 14.3.2 | Numbness (Safety Population) |
| Table 14.3.3.1 | Device deficiency per visit (Safety Population) |
| Table 14.3.3.2 | Device deficiency (number of events and subjects) (Safety Population) |

# 3.7.3 List of figures

| Table | Title |
|---|---|
| Figure 14.1.1 | Audiogram of Unaided Air Conduction and Bone Conduction, by Osia side and Non Osia side, and by masked and unmasked – Visit 1, Pre-Operative - SSD patients (Safety population) |
| Figure 14.1.2 | Audiogram of Unaided Air Conduction and Bone Conduction, by Osia side and Non Osia side, and by masked and unmasked – Visit 1, Pre-Operative - Conductive/Mixed hearing loss patients (Safety population) |
| Figure 14.2.1.1 | PTA4 - Free field Osia System vs Unaided (ITT Population) |
| Figure 14.2.1.2 | PTA4 - Free field Osia System vs Unaided (PP Population) |
| Figure 14.2.1.3 | PTA4 - Free field Osia System vs Unaided by Mixed/SSD (ITT Population) |
| Figure 14.2.1.4 | PTA4 - Free field Osia System vs Unaided by Mixed/SSD (PP Population) |
| Figure 14.2.1.5 | PTA4 - Free field Osia System vs Aided Softband (ITT Population) |
| Figure 14.2.1.6 | PTA4 - Free field Osia System vs Aided Softband (PP Population) |
| Figure 14.2.1.7 | PTA4 - Free field Osia System vs Aided Softband by Mixed/SSD (ITT Population) |
| Figure 14.2.1.8 | PTA4 - Free field Osia System vs Aided Softband by Mixed/SSD (PP Population) |
| Figure 14.2.2.1 | SNR - Free field Osia System vs Unaided (ITT Population) |
| Figure 14.2.2.2 | SNR - Free field Osia System vs Unaided (PP Population) |
| Figure 14.2.2.3 | SNR - Free field Osia System vs Unaided by Mixed/SSD (ITT Population) |
| Figure 14.2.2.4 | SNR - Free field Osia System vs Unaided by Mixed/SSD (PP Population) |
| Figure 14.2.2.5 | SNR - Free field Osia System vs Aided Softband (ITT Population) |
| Figure 14.2.2.6 | SNR - Free field Osia System vs Aided Softband (PP Population) |
| Figure 14.2.2.7 | SNR - Free field Osia System vs Aided Softband by Mixed/SSD (ITT Population) |

| | 33 |
|---|---|
| Figure 14.2.2.8 | SNR - Free field Osia System vs Aided Softband by Mixed/SSD (PP Population) |
| Figure 14.2.3.1 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB (ITT Population) |
| Figure 14.2.3.2 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB (PP Population) |
| Figure 14.2.3.3 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB by Mixed/SSD (ITT Population) |
| Figure 14.2.3.4 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB by Mixed/SSD (PP Population) |
| Figure 14.2.3.5 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB vs Aided Softband (ITT Population) |
| Figure 14.2.3.6 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB vs Aided Softband (PP Population) |
| Figure 14.2.3.7 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB vs<br>Aided Softband by Mixed/SSD (ITT Population) |
| Figure 14.2.3.8 | Adaptive speech recognition in Speech in Quiet for 50, 65 and 80 dB vs<br>Aided Softband by Mixed/SSD (PP Population) |

# 4 REFERENCES

### 4.1 Internal References

| ID | Document Title | Number |
|----|----------------|--------|

# 4.2 External References

| ID | Document Title | Number |
|----|----------------|--------|

# 5 CHANGE HISTORY

| Version | Change | Author | Date |
|---------|--------------------------|--------|-----------|
| 1.0 | Introduction of document | | 26-MAR-20 |

# **6** DEFINITIONS

| Term | Description |
|-------|--------------------------------------------|
| APHAB | Abbreviated Profile of Hearing Aid Benefit |
| BCHI | Bone conduction hearing implant |



| Term | Description |
|---|---|
| CHL | Conductive Hearing Loss |
| dB | Decibel |
| DLC | Digital Link Calibration |
| HUI | Health Utilities Index |
| Hz | Hertz |
| ITT | Intention to treat |
| Max | Maximum |
| MHL | Mixed Hearing Loss |
| Min | Minimum |
| n | Number |
| OSI | Active Osseointegrated Steady-State Implant System |
| PP | Per protocol |
| PTA4 | Pure Tone Average for and (mean of 500, 1000, 2000 and 4000Hz). Different definitions for audiogram on MHL/CHL/SSD patients. |
| SD | Standard deviation |
| SEM | Standard error of the mean |
| SNR | Speech to noise ratio |
| SSD | Single sided deafness |
| SSQ | Speech, Spatial and Qualities of Hearing Scale |